CLINICAL TRIAL: NCT01895140
Title: A Pragmatic Randomized Clinical Evaluation of Renal Denervation for Treatment Resistant Hypertension
Brief Title: A Study of Renal Denervation in Patients With Treatment Resistant Hypertension
Acronym: PaCE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Manufacturer updated device technology.
Sponsor: Dr. Harindra Wijeysundera (Other)
Collaborators: Medtronic (Industry); Mars Excellence in Clinical Innovation and Technology Evaluation (Other)
Responsible Party: Sponsor-Investigator, Dr. Harindra Wijeysundera, Interventional Cardiologist, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 322-2012
Record Dates: First submitted 2013-06-26; First posted 2013-07-10 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Treatment-Resistant Hypertension
Keywords: Treatment-resistant hypertension; Renal denervation; Ambulatory blood pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early renal denervation (Experimental): Renal denervation takes place immediately after patient is randomized.
  Interventions: Device: Renal denervation device
- Delayed renal denervation (Other): Renal denervation takes place 6 months after the patient is randomized.
  Interventions: Device: Renal denervation device

INTERVENTIONS:
Device: Renal denervation device
  Other Names: Medtronic Symplicity™ Catheter Device

SUMMARY:
The purpose of this study is to evaluate the clinical and economic impact of implementation of renal denervation with the Symplicity™ Catheter System for treatment-resistant hypertension in Ontario, Canada.

DETAILED DESCRIPTION:
This is a pragmatic randomized trial of renal nerve denervation for treatment resistant hypertension. This is part of a ministry sponsored MaRS-EXCITE program, to conduct early market health technology assessment, in order to determine appropriateness for provincial funding. We will assess the effectiveness, safety, economic attractiveness and feasibility of implementation of renal nerve denervation for treatment resistant hypertension. This will involve a new model of care which will include a multi-disciplinary team approach to these patients. Treatment resistant hypertension is defined as patients with uncontrolled hypertension despite being on optimal doses of 3 or more anti-hypertensive medications. Patients will be randomized to either standard treatment or renal nerve denervation and followed for 6 months to determine impact on blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Ontario residents
* Aged 18 and over
* Diagnosis of treatment-resistant hypertension after assessment and optimization by a hypertension specialist following recommended evaluation and diagnosis as outlined by the American Heart Association
* Office systolic blood pressure ≥ 160 mmHg (≥ 150 mmHg for patients with type II diabetes mellitus) prior to optimization by a hypertension specialist
* Baseline average systolic 24 hour ambulatory blood pressure of ≥ 135 mmHg after optimization and prior to randomization
* Prescribed 3 or more antihypertensive medications of different classes, both prior to optimization and at randomization, one of which must be a diuretic (a medication can be counted more than once if it acts on different receptors)
* Suitable renal artery anatomy based on CT/MRI/renal angiography imaging: both renal arteries > 20 mm in length and > 4 mm in diameter without significant fibromuscular disease or renal artery stenosis (>50%)

Exclusion Criteria:

* Secondary causes of hypertension:

  1. Primary aldosteronism (secondary to adrenal adenoma)
  2. Chronic kidney disease: creatinine clearance or eGFR < 45 ml/min/1.73m² (measured on 24 hour urine preferably or MDRD)
  3. Pheochromocytoma
  4. Cushing's syndrome
  5. Aortic coarctation (differential in brachial or femoral pulses, systolic bruit)
* Type 1 diabetes mellitus
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Average systolic 24-hour ambulatory blood pressure | 6 months

SECONDARY OUTCOMES:
Proportion of patients achieving target systolic blood pressure (on average 24-hour ambulatory blood pressure of <130 mmHg) on the same or fewer medications at the time of randomization | 6 months
Average daytime and average night-time systolic ambulatory blood pressure | 6 months
Variability of 24-hour ambulatory systolic blood pressure | 6 months
Average office blood pressure using an approved, automated office blood pressure device | 6 months
Hypertensive medication complexity index (MRCI) | 6 months
Number of hypertensive medications | 6 months
Peri-procedural mean cost per patient in Canadian dollars | 12 months
Generic quality of life (EQ-5D) | 6 months
Body Mass Index (BMI) | 6 months
24-hour urine sodium | 6 months
Acute periprocedural renal injury | 72 hours post procedure
Creatinine clearance measured on 24-hour urine (% change from baseline & indexed to Body Surface Area) | 6 months
Vascular complications (dissection, pseudoaneurysm, AV fistula) | 6 months
Evidence of renal artery stenosis compared to pre-procedure (determined by renal imaging, CT or MRA) for early intervention group | 6 months
Composite cardiovascular endpoints (fatal & non-fatal MI, new onset heart failure, stroke, beginning dialysis, hospitalization for cardiovascular/renal reasons, increase in hypertension medications) | 6 months
Microalbumin to creatinine ratio (MACR) from random urine sample (% change from baseline) | 6 months
24-hour urine sodium (% change from baseline) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Harindra C. Wijeysundera, MD, Principal Investigator — Sunnybrook Research Institute
Locations (2):
- Canada (2):
  - Sunnybrook Research Institute, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario